CLINICAL TRIAL: NCT03536260
Title: Evaluation of Marginal Bone Loss After Immediate Implant Placement in Maxillary Esthetic Zone With Nanobone Versus Xenograft (Randomized Clinical Trial)
Brief Title: Evaluation of Marginal Bone Loss After Immediate Implant Placement in Maxillary Esthetic Zone With Nanobone Versus Xenograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdullah Mohammed Farahat, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FarahatMBL
Record Dates: First submitted 2018-04-05; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Implant Placement in Maxillary Esthetic Zone
MeSH Terms: interventions — Mutagenesis, Insertional; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant with Xenograft (Active Comparator)
  Interventions: Device: Implant with Xenograft
- Immediate implant with Nanobone (Active Comparator)
  Interventions: Device: Implant with NanoBone graft

INTERVENTIONS:
Device: Implant with NanoBone graft — Using of NanoBone graft to fill the gap in the socket after immediate implant placement
  Arms: Immediate implant with Nanobone
Device: Implant with Xenograft — Using of Xenograft to fill the gap in the socket after immediate implant placement
  Arms: Immediate implant with Xenograft

SUMMARY:
Immediate implant placement has a success rate from 94-100 % . After tooth extraction there is a loss in the horizontal and vertical dimension by about 3-6 mm and 1-2 mm respectively and alveolar crest resorption of about 44% especially through 6 months after extraction.

After immediate implant placement there is usually a void between the implant and the socket walls which is called jumping distance or gap which may heal spontaneously or need bone graft to bridge the space. If the gap is 1-2 mm it may heal spontaneously more than that this will need bone graft. There is no evidence that the graft impairs osseointegration Development of artificial bone has increasingly progressed in the last few years. Nanobone "nanocrystalline hydroxyapatite embedded in a porous silica gel matrix bone graft is introduced which has osseoconductive and biomimetic properties .the sub-micron modification in the bone substitute will enhance osteogenic property. It bind to the bone by stimulation of osteoblast activity and enhance growth factors which improve bone healing and provide more strength and stability to the implant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth in upper esthetic zone indicated for extraction, presence of at least 4 mm of bone beyond the root apex to guarantee implant primary stability, implant placement within the alveoli confines.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony Walls after extraction.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Crestal Bone Loss in grafted socket | 3 months after implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided